CLINICAL TRIAL: NCT06169475
Title: Effect of Dexmedetomidine vs Esmolol or Placebo on Cerebral Hemodynamics in Septic Shock: A Randomized Clinical Trial.
Brief Title: Effect of Dexmedetomidine vs Esmolol or Placebo on Cerebral Hemodynamics in Septic Shock
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xinchen Wang (Other)
Collaborators: Tibet Autonomous Region People's Hospital (Other)
Responsible Party: Sponsor-Investigator, Xinchen Wang, Attending Doctor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D-E-P-sepsis
Record Dates: First submitted 2023-11-27; First posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Septic Shock; Stress Response; Cerebral Hemodynamics
Keywords: Septic shock; Stress response; Trans-cranial Doppler
MeSH Terms: conditions — Shock, Septic; Fractures, Stress | interventions — Dexmedetomidine; esmolol

STUDY DESIGN:
Who Masked: Participant
Masking Description: The participants who under deep sedation are blinded to the grouping.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- dexmedetomidine group (Experimental)
  Interventions: Drug: Dexmedetomidine Hydrochloride
- esmolol group (Experimental)
  Interventions: Drug: Esmolol Hydrochloride
- control group (No Intervention)

INTERVENTIONS:
Drug: Dexmedetomidine Hydrochloride — The continuous intravenous infusion of dexmedetomidine (0.1mg/ml) will start at 0.1ug/kg/h, increasing every 20 minutes by a step change of 0.05-0.2ug/kg/h to reach the target heart rate with the expectation that this should be within 12 hours. The infusion will be reduced by step change, and if necessary, ultimately stopped if the heart rate fall below 80b.p.m..
  Arms: dexmedetomidine group
Drug: Esmolol Hydrochloride — The continuous intravenous infusion of esmolol (10mg/ml) will start at 20mg/h, increasing every 20 minutes by a step change of 20mg/h to reach the target heart rate with the expectation that this should be within 12 hours. The infusion will be reduced by step change, and if necessary, ultimately stop if the heart rate fall below 80b.p.m..
  Arms: esmolol group

SUMMARY:
Sepsis is defined as life-threatening organ dysfunction caused by a dysregulated host response to infection. Some researchers proposed that the dysregulated response or organ dysfunction can be lessened by reducing the stress response, which further reduce complication and mortality rates of sepsis. Dexmedetomidine is alpha adrenergic receptor agonist, presenting sympatholytic action in certain parts of the brain with anxiolytic, sedative, and pain killing effects. In the experiments of sepsis animal model, dexmedetomidine have been proved to improve serum lactate clearance and the microcirculation. Dexmedetomidine may inhibit inflammation, as it enhances the activity of the immune system while reducing its systemic reaction and lowering cytokine concentrations. There are also evidences in clinical trials with definite safety that dexmedetomidine reduced inflammation, reduced vasopressor requirements and improved organ function. The beta antagonist esmolol has been proposed as a therapy to lower heart rate, thereby improving diastolic filling time, and improving cardiac output, resulting in a reduction in vasopressor support. A recent meta-analysis of 8 randomized studies using esmolol suggested that the 32% risk ratio decreased 28-day mortality, and a meta-analysis of 7 studies using esmolol in patients with sepsis and septic shock was associated with 32% lower 28-day mortality. However, the effect of anti-stress drugs on cerebral hemodynamics is unknown. In this study, investigators are going to apply the technique of transcranial Doppler to assess the reaction of cerebral blood flow in anti-stress group and control group.

DETAILED DESCRIPTION:
It is a single-blinded, single-center, randomized trial. Patients with septic shock established within 24 hours in the ICU of Tibet Autonomous Region People's Hospital will be screened for recruitment. After adequate fluid resuscitation, continuous infusion of norepinephrine is given to the patients to maintain a mean arterial pressure (MAP) of 65-75 millimeter of mercury (mmHg). Midazolam and fentanyl are given to achieve the goal sedation of bispectral index (BIS) 40-60, patients who are still with tachycardia (heart rate over 100 b.p.m.) will be recruited. After recruitment, patients in accordance with the random number table are divided into dexmedetomidine group, esmolol group and control group (T0). Patients in the two experimental groups are required to achieve the heart rate goal of 75-95 b.p.m. in one hour by adjusting the dose of dexmedetomidine or esmolol every twenty minutes. All patients acquired the hemodynamic evaluation at T1, T2, T3, T4 (6, 12, 18, 24hours after enrollment). The hemodynamic evaluation including transcranial Doppler of middle cerebral artery(MCA), deep middle cerebral vein (DMCV), basal vein Rosenthal (BVR) and transverse sinus (TS), hemodynamic parameters acquired by the pressure-recording analytical method through peripheral arterial with Mostcare. Demographic characteristics, diagnosis, laboratory reports and drug dose are collected during the study.

ELIGIBILITY:
Inclusion Criteria:

1. 18 ~ 80 years old.
2. Patients established septic shock according to sepsis 3.0 criteria.
3. Under deep sedation of BIS 40-60 with midazolam and fentanyl.
4. After achieving the goal sedation, patients are still with tachycardia (heart rate over 100 b.p.m..

Exclusion Criteria:

1. Pregnancy.
2. Patients with severe arrhythmia.
3. Patients with aortic or aortic valve disease.
4. Patients with mechanical circulatory assist device (e.g. extracorporeal membrane oxygenation (ECMO), intra-aortic balloon pump (IABP), etc).
5. Patients with cerebral trauma.
6. Any contraindication to the use of transcranial doppler.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
The cerebral hemodynamic change caused by the anti-stress therapy | Hour 0, Hour 6, Hour 12, Hour 18 and Hour 24.
  The cerebral hemodynamics will be evaluated according to the features of the blood flow of MCA, DMCV, BVR and TS measured by transcranial doppler, as well as regional cerebral oxygen saturation measured by the near infrared spectroscopy at Hour 0, Hour 6, Hour 12, Hour 18 and Hour 24. The difference will be acquired by contrasting between two intervention group and one control group.

SECONDARY OUTCOMES:
The systemic hemodynamic change caused by anti-stress therapy | Hour 0, Hour 6, Hour 12, Hour 18 and Hour 24
  The systemic hemodynamic changes will be acquired through the pressure-recording analytical method with Mostcare, blood pressure and electro cardiac monitor, central venous pressure (CVP) monitor, trans thoracic echocardiography, and blood gas at Hour 0, Hour 6, Hour 12, Hour 18 and Hour 24. The difference will be acquired by contrasting between two intervention group and one control group

CONTACTS AND LOCATIONS:
Overall Officials: Wei Du, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Chinese Academy of Medical Science, Beijing, China

REFERENCES:
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Du W, Liu D, Long Y, Wang X. The beta-Blocker Esmolol Restores the Vascular Waterfall Phenomenon After Acute Endotoxemia. Crit Care Med. 2017 Dec;45(12):e1247-e1253. doi: 10.1097/CCM.0000000000002721. PMID 28991824
- [Background] Dardalas I, Stamoula E, Rigopoulos P, Malliou F, Tsaousi G, Aidoni Z, Grosomanidis V, Milonas A, Papazisis G, Kouvelas D, Pourzitaki C. Dexmedetomidine effects in different experimental sepsis in vivo models. Eur J Pharmacol. 2019 Aug 5;856:172401. doi: 10.1016/j.ejphar.2019.05.030. Epub 2019 May 17. PMID 31108055
- [Background] Ohta Y, Miyamoto K, Kawazoe Y, Yamamura H, Morimoto T. Effect of dexmedetomidine on inflammation in patients with sepsis requiring mechanical ventilation: a sub-analysis of a multicenter randomized clinical trial. Crit Care. 2020 Aug 10;24(1):493. doi: 10.1186/s13054-020-03207-8. PMID 32778146
- [Background] Scibelli G, Maio L, Sasso M, Lanza A, Savoia G. Dexmedetomidine: Current Role in Burn ICU. Transl Med UniSa. 2017 Jul 1;16:1-10. eCollection 2017 Jan. PMID 28775963
- [Background] Nakashima T, Miyamoto K, Shima N, Kato S, Kawazoe Y, Ohta Y, Morimoto T, Yamamura H; DESIRE Trial Investigators. Dexmedetomidine improved renal function in patients with severe sepsis: an exploratory analysis of a randomized controlled trial. J Intensive Care. 2020 Jan 2;8:1. doi: 10.1186/s40560-019-0415-z. eCollection 2020. PMID 31908779
- [Background] Zhang J, Chen C, Liu Y, Yang Y, Yang X, Yang J. Benefits of esmolol in adults with sepsis and septic shock: An updated meta-analysis of randomized controlled trials. Medicine (Baltimore). 2022 Jul 8;101(27):e29820. doi: 10.1097/MD.0000000000029820. PMID 35801730